CLINICAL TRIAL: NCT03578380
Title: Supermicrosurgery for Breast Cancer Survivors With Lymphedema. -Prospective Randomized Clinical and Patient-reported Outcomes.
Brief Title: Supermicrosurgery for Breast Cancer Survivors With Lymphedema.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: University of Oslo (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prosjektnr 1097.19
Record Dates: First submitted 2017-06-12; First posted 2018-07-06 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-12

CONDITIONS: Secondary Lymphedema; Breast Cancer
Keywords: Lymphovenous bypass; Lymphovenous anastomosis; Supermicrosurgery; Lymphangiography; MD Anderson Lymphedema Stage
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery (Experimental): Lymphovenous anastomosis
  Interventions: Procedure: Surgery
- Compression (Active Comparator): Conservative treatment with physiotherapy and compression
  Interventions: Other: Compression and drainage therapy

INTERVENTIONS:
Procedure: Surgery — Lymphovenous anastomosis
  Arms: Surgery
Other: Compression and drainage therapy — Treatment with compression stockings and manual drainage (massage therapy)
  Arms: Compression

SUMMARY:
A randomised prospective investigation of volume and quality of life results with lymphovenous anastomosis in patients with unilateral arm lymphedema after breast cancer using Indocyanine Green lymphangiography and MD Anderson Staging.

DETAILED DESCRIPTION:
This is a randomized study comparing lymphovenous anastomosis versus conservative (compression) treatment for lymphoedema after breast cancer surgery - 50 patients to be included in each study arm. The primary endpoint is volume change measured by submersion and changes in arm circumference at defined levels from the wrist. Secondary endpoint is health related quality of life measured by questionnaire Short Form 36 (SF-36), Hospital Anxiety Depression Score (HADS), Fatigue Questionnaire (FQ) and a disease-specific questionnaire, Upper Limb Lymphedema score (ULL27).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lymphedema of the arm secondary to breast cancer treatment. Stage 1-3 operable lymphedema.

Exclusion Criteria:

* Frequent or severe cellulitis. All other lymphedema.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Volume | 12 months
  Volume of arm as described by submersion and circumference measures

SECONDARY OUTCOMES:
Health related quality of life ULL27 | 12 months
  To be measured by questionnaire "Upper Limb Lymphedema score 27" (ULL27) by Professor Robert Launois at REES France. The scale measures health related quality of life in patients with upper limb lymphedema.
  Construction: 27 questions rated from 1 (lowest quality of life) to 5 highest quality of life.
  Dimensions: There are 3 dimensions assessing symptoms, self value, everyday social life. Total score 27-135 Symptom score: 18-90 Self value: 5-25 Social life: 4-20 Question 20 and 22 are part of the self value dimension and are control questions with reverse scores, i.e 1 represents highest quality of life and 5 represents lowest quality of life. The scores for question 20 and 22 are later reversed when adding the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Johan Sandberg, MD, Principal Investigator — Sykehuset Telemark
Locations (1):
- Sykehuset Telemark, Skien, Telemark, Norway

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers